CLINICAL TRIAL: NCT02234297
Title: A Phase 1 Dose Escalation/Expansion Study of BLZ-100 Administered by Intravenous Injection in Adult Subjects With Glioma Undergoing Surgery
Brief Title: Safety Study of BLZ-100 in Adult Subjects With Glioma Undergoing Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Blaze Bioscience Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: BB-002
Record Dates: First submitted 2014-08-04; First posted 2014-09-09 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Glioma
Keywords: Glioma; Tumor Paint; BLZ100
MeSH Terms: conditions — Glioma | interventions — tozuleristide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BLZ-100 (Experimental)
  Interventions: Drug: BLZ-100

INTERVENTIONS:
Drug: BLZ-100
  Other Names: Tumor Paint

SUMMARY:
Many types of cancer are primarily treated with surgery and patient survival is directly related to the extent to which the tumor is able to be removed. It is often difficult for surgeons to distinguish tumor tissue from normal tissue or to detect tumor cells that have spread from the original tumor site, resulting in incomplete removal of the tumor and reduced patient survival. In some sites, such as the brain, it is critical to avoid damage to normal tissue around the tumor to prevent adverse effects of surgery on function. We hypothesize that BLZ-100 will improve surgical outcomes by allowing surgeons to visualize the edges of the tumor and small groups of cancer cells that have spread to other sites in real-time as operate. This is a safety study to assess the safety of BLZ-100 in patients with gliomas undergoing surgery.

DETAILED DESCRIPTION:
Subjects who provide voluntary written informed consent will be screened for eligibility. Subjects meeting all of the inclusion and none of the exclusion criteria will be eligible to participate.

Subjects will be required to arrive at the hospital (or phase 1 unit if applicable) for dosing at least 2 hours before the planned surgical excision. Following dosing, subjects will be monitored for safety and surgical excision will occur at least 2 hours after study product administration.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18- 75 years.
2. Subjects must have glioma for which surgical resection is clinically indicated. Grade I, II, III and IV glioma patients will be included (for example glioblastoma, astrocytoma, and oligodendroglioma). Histological confirmation not required prior to surgery. Subjects with recurrent disease will be eligible only if the duration between last brain surgery and scheduled new surgery is ≥3 months. The grade of a recurrent tumor will be presumed that of the primary tumor for purposes of group allocation.
3. Able to provide written informed consent.
4. If of child-bearing potential, agree to the continued use of effective contraceptive from study entry (Informed consent) through 30 days after BLZ-100 administration.
5. Available for all study visits and able to comply with all study requirements

Exclusion Criteria:

1. Evidence of metastatic disease.
2. Female who is lactating/breastfeeding
3. Female with a positive pregnancy test or who is planning to become pregnant during the duration of the study.
4. Karnofsky Performance Status of <60%.
5. Any of the following laboratory abnormalities at Screening:

   1. Neutrophil count <1.5 x 10^9/L
   2. Platelets <75 x 10^9/L
   3. Hemoglobin <10 g/dL (may be determined following transfusion)
   4. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3x upper limit of normal (ULN)
   5. Total bilirubin >1.5x upper limit of reference range (unless Gilbert's syndrome or extrahepatic source as denoted by increased indirect bilirubin fraction)
   6. International Normalized Ratio (INR) >1.5
   7. Creatinine >1.5x ULN
6. Positive serology for human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis B virus (HBV).
7. QTc prolongation >450 msec
8. History of hypersensitivity or allergic reactions requiring corticosteroids, epinephrine and/or hospitalization.
9. Uncontrolled asthma or asthma requiring oral corticosteroids.
10. Known or suspected sensitivity to MRI contrast agents or excipients in the study drug product.
11. Known or suspected sensitivity to Indocyanine green (ICG).
12. Unstable angina, myocardial infarction, known or suspected transient ischemic events or stroke within 24 weeks of start of Screening.
13. Uncontrolled hypertension.
14. Receipt of photosensitizing drugs within 30 days of Screening.
15. Any ongoing medications which might generate fluorescence or according to label, might generate a photochemical reaction. These include haematoporphyrin derivatives and purified fractions; Photofrin®; and the precursors of protoporphyrin IX (5-Aminolevulinic acid) used in Gliolan or Hexvix.
16. Received an investigational drug or device within 30 days of enrollment.
17. Prior treatment with BLZ-100.
18. Any concurrent condition, including psychological and social situations, which, in the opinion of the investigator, would impact adversely on the subject or the interpretation of the study data.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-10; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Seven days after study drug administration
  Safety will be assessed by physical examination and measurement of vital signs and laboratory safety parameters.

SECONDARY OUTCOMES:
Change in concentration of BLZ-100 in the blood | Prior to dosing and at 1 minute, 5 minutes, 15 mins, 30 mins, 60 mins and 120 mins after end of injection
  BLZ-100 levels in blood will be analyzed by chemical means and these data will be used to calculate pharmacokinetic parameters.

OTHER OUTCOMES:
Fluoresence signal in excised brain tumor and normal brain cancer | at least 2 hours post-dose
  Fluorescence signal in sections of excised tumor and adjacent normal tissue will be measured using an infrared imaging system.

CONTACTS AND LOCATIONS:
Overall Officials: Chirag Patil, Principal Investigator — Cedars-Sinai Medical Center
Locations (2):
- Cedars-Sinai Medical Center, Los Angeles, California, United States
- NEWRO Foundation, Brisbane, Queensland, Australia